CLINICAL TRIAL: NCT04489056
Title: The Human Microbiome in pPROM, Preterm Birth and the Neonatal Infant: a Prospective Longitudinal Pilot-study
Brief Title: Microbiome in Preterm Birth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: University of Vienna (Other)
Responsible Party: Principal Investigator, Alex Farr, MD PhD, Prof. Alex Farr, MD PhD, Medical University of Vienna
Other Study IDs: 1668/2020
Record Dates: First submitted 2020-07-20; First posted 2020-07-28 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Vaginal Microbiome
Keywords: Vaginal microbiome; Preterm birth; Neonatal microbiome
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Analysis of the maternal vaginal, rectal, placental and uterus microbiome Analysis of the neonatal buccal, skin and stool micro biome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: This group will consist of 50 pregnant women, who experienced pPROM between 22+5 and 28+0 gestational weeks, either presenting at the primary study site, or being referred from other hospitals, and delivered at preterm by cesarean section.
  Interventions: Genetic: Swabs for microbiome analysis
- Control group: This group will consist of 50 pregnant women, who are scheduled for elective cesarean section at the outpatient department of the primary study site, between a 32+0 and 37+0 gestational weeks, and delivered at term by cesarean section.
  Interventions: Genetic: Swabs for microbiome analysis

INTERVENTIONS:
Genetic: Swabs for microbiome analysis — After informed consent, vaginal swabs will be collected during speculum examination from the lateral vaginal wall and posterior fornix vaginae using a sterile cotton swab combined with an epithelial brush. A rectal swab will be collected by insertion of a sterile swab into the anal sphincter. Intraoperative swabs of the placenta and uterine cavity will be collected during caesarean section under sterile conditions. Neonatal swabs (buccal mucosa and skin) will be collected directly after delivery and in the neonatal period. Stool samples will be taken from the meconium, defined as first stool of the infant and the stool of the newborn in the neonatal period.

SUMMARY:
The aims of this prospective longitudinal case-control pilot-study are (1) to characterize the changes of the vaginal, uterine and placental microbiome in pregnant women experiencing pPROM with immediate hospitalization and consecutive caesarean section at preterm, in comparison to uneventful term births with elective cesarean section, as well as (2) to evaluate the influence of the maternal on the neonatal microbiome and the early neonatal outcome in pPROM preterm cases, in comparison to uneventful term births.

The first aim will be achieved by collecting vaginal and rectal swabs for microbiome analysis in women experiencing pPROM, followed by uterine and placental swabs that are collected during the caesarean section. Control samples will be collected at the same time points from women undergoing elective caesarean section at term. The second aim will be achieved by microbiome analysis of rectal, oral/buccal, and skin swabs taken from newborns that are either born preterm after pPROM, or at term, both by caesarean section.

DETAILED DESCRIPTION:
A total of 100 study participants will be included, assigned to one of the following groups:

Study group:

• This group will consist of 50 pregnant women, who experienced pPROM between 22+5 and 28+0 gestational weeks, either presenting at the primary study site, or being referred from other hospitals, and delivered at preterm by cesarean section.

Control group:

• This group will consist of 50 pregnant women, who are scheduled for elective cesarean section at the outpatient department of the primary study site, between a 32+0 and 37+0 gestational weeks, and delivered at term by cesarean section.

Recruitment:

Recruitment of all patients will take place at the Medical University of Vienna, Department of Obstetrics and Gynecology. Women in the study group will be referred from outside hospitals or will present for any reason at our department. Verification of pPROM will be performed by speculum examination and detection of amniotic fluid pooling. In case of unclear findings, an enzymatic test (e.g., Amnisure®, QUIAGEN Sciences, LLC; Germantown, MD 20874, USA) will be conducted. Following pPROM verification, women who meet the inclusion criteria will be offered to participate in the study. Those who experience a spontaneous vaginal delivery instead of a cesarean section due to any reason, will be considered as drop-out. Women in the control group will be recruited during their routine presentation for elective cesarean section (for any reason that does not meet the exclusion criteria of the study) that will be scheduled at term. Those who experience preterm birth although being scheduled for elective cesarean at term, will be considered as drop-out. During their consultation at the outpatient department, these women will be offered to participate in the study.

Sampling:

All swabs will be collected from sub-investigators of this study using a standardized procedure. For anonymization, only the collection time point, location and ward will be marked on the swab tubes. After informed consent, vaginal swabs will be collected during speculum examination from the lateral vaginal wall and posterior fornix vaginae using a sterile cotton swab combined with an epithelial brush. A rectal swab will be collected by insertion of a sterile swab into the anal sphincter. Intraoperative swabs of the placenta and uterine cavity will be collected during caesarean section under sterile conditions. Neonatal swabs (buccal mucosa and skin) will be collected directly after delivery and in the neonatal period. Stool samples will be taken from the meconium, defined as first stool of the infant and the stool of the newborn in the neonatal period. All specimens will immediately be stored at -80°C after collection. The epithelial brush will be put into RNAlater® RNA stabilization solution and stored at -80°C.

Microbiome analysis:

Microbiome analysis will be performed at the Joint Microbiome Facility (JMF) of the Medical University of Vienna and the University of Vienna. Testing will be performed by sub- investigators at the JMF. The microbial community composition in collected stool swab samples will be determined by 16S rRNA gene amplicon sequencing. Briefly, DNA will be extracted with the QIAamp Microbiome Kit or QIAamp DNA Mini Kit (for swab and stool samples, respectively), followed by 16S rRNA gene amplification and barcoding as previously described. Multiplexed amplicon samples sequenced on the Illumina MiSeq platform at the JMF. Negative controls performed during DNA extraction and 16S rRNA gene amplification are routinely included in the sample processing workflow. The obtained sequence data will be quality-filtered and demultiplexed, followed by amplicon sequencing variant (ASV) inference with DADA2,16 enabling analysis at the highest possible taxonomic resolution. Resulting ASV sequences will be taxonomically classified using SINA with the newest release of the the SILVA SSU rRNA database. If necessary, contaminants will be removed in silico using the decontam software package.

Perinatal data:

In addition to swab sampling and analysis, the following perinatal parameters will be collected, using the PIA Fetal Database, version 5.6.16.917 (GE Viewpoint, Munich, Germany): Maternal age [number], parity [number], tertiary education [yes/no], ethnicity [category], relationship status [category], body mass index [number], nicotine abuse [yes/no], history of pPROM [yes/no], history of PTB [yes/no], preexisting diseases [category], vaginal infection screening [yes/no], cervical insufficiency [yes/no], preeclampsia [yes/no], bleeding [yes/no], antenatal steroid prophylaxis [yes/no], ongoing antibiotic treatment [yes/no], tocolysis [yes/no], magnesium prophylaxis [yes/no], gestational week at delivery [number], birthweight [number], Apgar score at 1/5/10 minutes [number], umbilical cord arterial pH [number], transfer to neonatal intensive care unit [yes/no].

ELIGIBILITY:
Inclusion Criteria:

* Maternal age ≥18 years at the time of study enrollment
* Singleton pregnancy
* Signed informed consent
* Confirmed preterm premature rupture of membranes (pPROM) or elective cesarean section for term birth (depending on study group)
* Gestational age at the time of pPROM between 22+5 and 28+0 weeks or ≥37+0 gestational weeks at the time of term cesarean section (depending on study group)

Exclusion Criteria:

* Maternal age <18 years at the time of study enrollment
* Multiple pregnancy
* Inability to consent to the participation in the study
* Ongoing antibiotic treatment or antibiotic treatment ≤2 weeks before study enrollment
* Vaginal sexual intercourse within 48 hours before study enrollment
* Fresh vaginal bleeding within 48 hours before study enrollment
* Maternal Hepatitis-B or Hepatitis-C infection (i.e., positive on PCR)
* Maternal HIV-infection (i.e., positive on PCR)
* Maternal diabetes mellitus or gestational diabetes

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: A total of 100 study participants, meeting all inclusion and non exclusion criteria, will be included, assigned to one of the following groups:
  Study group:
  • This group will consist of 50 pregnant women, who experienced pPROM between 22+5 and 28+0 gestational weeks, either presenting at the primary study site, or being referred from other hospitals, and delivered at preterm by cesarean section.
  Control group:
  • This group will consist of 50 pregnant women, who are scheduled for elective cesarean section at the outpatient department of the primary study site, between a 32+0 and 37+0 gestational weeks, and delivered at term by cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Changes of the vaginal microbiome after pPROM in comparison to term births | Till July 2021
  Abundance measurements (counts) of the amplicon sequence variants (ASVs), as well as ASV sum counts at higher taxonomic levels will be evaluated, to test for significant overlap or differences in microbial community composition in different sample groups. These parameters will be analyzed within each of the study groups, including longitudinal analyses to detect a potential difference from the onset of pPROM to the time of delivery or later (study group), or from pregnancy to the time of delivery or later (control group). In addition, ASVs and ASV sum counts will be compared between the study and control group at predetermined time points. Detection of significantly more abundant amplicon sequence variants between groups will be performed, and adjusted P-values will be calculated using the Benjamini-Hochberg method and differences supported with P- values <0.05 will be considered significant.
Changes of the rectal microbiome after pPROM in comparison to term births | Till July 2021
  Abundance measurements (counts) of the amplicon sequence variants (ASVs), as well as ASV sum counts at higher taxonomic levels will be evaluated, to test for significant overlap or differences in microbial community composition in different sample groups. These parameters will be analyzed within each of the study groups, including longitudinal analyses to detect a potential difference from the onset of pPROM to the time of delivery or later (study group), or from pregnancy to the time of delivery or later (control group). In addition, ASVs and ASV sum counts will be compared between the study and control group at predetermined time points. Detection of significantly more abundant amplicon sequence variants between groups will be performed, and adjusted P-values will be calculated using the Benjamini-Hochberg method and differences supported with P- values <0.05 will be considered significant.
Changes of the placental microbiome after pPROM in comparison to term births | Till July 2021
  Abundance measurements (counts) of the amplicon sequence variants (ASVs), as well as ASV sum counts at higher taxonomic levels will be evaluated, to test for significant overlap or differences in microbial community composition in different sample groups. These parameters will be analyzed within each of the study groups, including longitudinal analyses to detect a potential difference from the onset of pPROM to the time of delivery or later (study group), or from pregnancy to the time of delivery or later (control group). In addition, ASVs and ASV sum counts will be compared between the study and control group at predetermined time points. Detection of significantly more abundant amplicon sequence variants between groups will be performed, and adjusted P-values will be calculated using the Benjamini-Hochberg method and differences supported with P- values <0.05 will be considered significant.
Changes of the uterine microbiome after pPROM in comparison to term births | Till July 2021
  Abundance measurements (counts) of the amplicon sequence variants (ASVs), as well as ASV sum counts at higher taxonomic levels will be evaluated, to test for significant overlap or differences in microbial community composition in different sample groups. These parameters will be analyzed within each of the study groups, including longitudinal analyses to detect a potential difference from the onset of pPROM to the time of delivery or later (study group), or from pregnancy to the time of delivery or later (control group). In addition, ASVs and ASV sum counts will be compared between the study and control group at predetermined time points. Detection of significantly more abundant amplicon sequence variants between groups will be performed, and adjusted P-values will be calculated using the Benjamini-Hochberg method and differences supported with P- values <0.05 will be considered significant.
Changes of the neonatal microbiome of neonates born after pPROM in comparison to neonates experiencing a term birth | Till July 2021
  Abundance measurements (counts) of the amplicon sequence variants (ASVs), as well as ASV sum counts at higher taxonomic levels will be evaluated, to test for significant overlap or differences in microbial community composition in different sample groups. These parameters will be analyzed within each of the study groups, including longitudinal analyses to detect a potential difference from the onset of pPROM to the time of delivery or later (study group), or from pregnancy to the time of delivery or later (control group). In addition, ASVs and ASV sum counts will be compared between the study and control group at predetermined time points. Detection of significantly more abundant amplicon sequence variants between groups will be performed, and adjusted P-values will be calculated using the Benjamini-Hochberg method and differences supported with P- values <0.05 will be considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Farr, MD PhD, Principal Investigator — Medical University of Vienna; Herbert Kiss, MD MBA, Study Chair — Medical University of Vienna; Angelika Berger, MD MBA, Study Chair — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Dept. of Obstetrics and Gynecology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data if required and in accordance with data protection regulations

REFERENCES:
- [Background] Chu DM, Seferovic M, Pace RM, Aagaard KM. The microbiome in preterm birth. Best Pract Res Clin Obstet Gynaecol. 2018 Oct;52:103-113. doi: 10.1016/j.bpobgyn.2018.03.006. Epub 2018 Apr 9. PMID 29753695
- [Background] Human Microbiome Project Consortium. Structure, function and diversity of the healthy human microbiome. Nature. 2012 Jun 13;486(7402):207-14. doi: 10.1038/nature11234. PMID 22699609
- [Background] Klindworth A, Pruesse E, Schweer T, Peplies J, Quast C, Horn M, Glockner FO. Evaluation of general 16S ribosomal RNA gene PCR primers for classical and next-generation sequencing-based diversity studies. Nucleic Acids Res. 2013 Jan 7;41(1):e1. doi: 10.1093/nar/gks808. Epub 2012 Aug 28. PMID 22933715
- [Background] Jovel J, Patterson J, Wang W, Hotte N, O'Keefe S, Mitchel T, Perry T, Kao D, Mason AL, Madsen KL, Wong GK. Characterization of the Gut Microbiome Using 16S or Shotgun Metagenomics. Front Microbiol. 2016 Apr 20;7:459. doi: 10.3389/fmicb.2016.00459. eCollection 2016. PMID 27148170
- [Background] Gosmann C, Anahtar MN, Handley SA, Farcasanu M, Abu-Ali G, Bowman BA, Padavattan N, Desai C, Droit L, Moodley A, Dong M, Chen Y, Ismail N, Ndung'u T, Ghebremichael MS, Wesemann DR, Mitchell C, Dong KL, Huttenhower C, Walker BD, Virgin HW, Kwon DS. Lactobacillus-Deficient Cervicovaginal Bacterial Communities Are Associated with Increased HIV Acquisition in Young South African Women. Immunity. 2017 Jan 17;46(1):29-37. doi: 10.1016/j.immuni.2016.12.013. Epub 2017 Jan 10. PMID 28087240
- [Background] O'Hanlon DE, Moench TR, Cone RA. In vaginal fluid, bacteria associated with bacterial vaginosis can be suppressed with lactic acid but not hydrogen peroxide. BMC Infect Dis. 2011 Jul 19;11:200. doi: 10.1186/1471-2334-11-200. PMID 21771337
- [Background] Dominguez-Bello MG, Costello EK, Contreras M, Magris M, Hidalgo G, Fierer N, Knight R. Delivery mode shapes the acquisition and structure of the initial microbiota across multiple body habitats in newborns. Proc Natl Acad Sci U S A. 2010 Jun 29;107(26):11971-5. doi: 10.1073/pnas.1002601107. Epub 2010 Jun 21. PMID 20566857
- [Background] Callahan BJ, DiGiulio DB, Goltsman DSA, Sun CL, Costello EK, Jeganathan P, Biggio JR, Wong RJ, Druzin ML, Shaw GM, Stevenson DK, Holmes SP, Relman DA. Replication and refinement of a vaginal microbial signature of preterm birth in two racially distinct cohorts of US women. Proc Natl Acad Sci U S A. 2017 Sep 12;114(37):9966-9971. doi: 10.1073/pnas.1705899114. Epub 2017 Aug 28. PMID 28847941
- [Background] Brown RG, Al-Memar M, Marchesi JR, Lee YS, Smith A, Chan D, Lewis H, Kindinger L, Terzidou V, Bourne T, Bennett PR, MacIntyre DA. Establishment of vaginal microbiota composition in early pregnancy and its association with subsequent preterm prelabor rupture of the fetal membranes. Transl Res. 2019 May;207:30-43. doi: 10.1016/j.trsl.2018.12.005. Epub 2018 Dec 27. PMID 30633889
- [Background] Stout MJ, Zhou Y, Wylie KM, Tarr PI, Macones GA, Tuuli MG. Early pregnancy vaginal microbiome trends and preterm birth. Am J Obstet Gynecol. 2017 Sep;217(3):356.e1-356.e18. doi: 10.1016/j.ajog.2017.05.030. Epub 2017 May 23. PMID 28549981
- [Background] Thorsen J, Brejnrod A, Mortensen M, Rasmussen MA, Stokholm J, Al-Soud WA, Sorensen S, Bisgaard H, Waage J. Large-scale benchmarking reveals false discoveries and count transformation sensitivity in 16S rRNA gene amplicon data analysis methods used in microbiome studies. Microbiome. 2016 Nov 25;4(1):62. doi: 10.1186/s40168-016-0208-8. PMID 27884206
- [Background] Davis NM, Proctor DM, Holmes SP, Relman DA, Callahan BJ. Simple statistical identification and removal of contaminant sequences in marker-gene and metagenomics data. Microbiome. 2018 Dec 17;6(1):226. doi: 10.1186/s40168-018-0605-2. PMID 30558668
- [Background] Pruesse E, Peplies J, Glockner FO. SINA: accurate high-throughput multiple sequence alignment of ribosomal RNA genes. Bioinformatics. 2012 Jul 15;28(14):1823-9. doi: 10.1093/bioinformatics/bts252. Epub 2012 May 3. PMID 22556368
- [Background] Quast C, Pruesse E, Yilmaz P, Gerken J, Schweer T, Yarza P, Peplies J, Glockner FO. The SILVA ribosomal RNA gene database project: improved data processing and web-based tools. Nucleic Acids Res. 2013 Jan;41(Database issue):D590-6. doi: 10.1093/nar/gks1219. Epub 2012 Nov 28. PMID 23193283
- [Background] Callahan BJ, McMurdie PJ, Rosen MJ, Han AW, Johnson AJ, Holmes SP. DADA2: High-resolution sample inference from Illumina amplicon data. Nat Methods. 2016 Jul;13(7):581-3. doi: 10.1038/nmeth.3869. Epub 2016 May 23. PMID 27214047
- [Background] Herbold CW, Pelikan C, Kuzyk O, Hausmann B, Angel R, Berry D, Loy A. Corrigendum: A flexible and economical barcoding approach for highly multiplexed amplicon sequencing of diverse target genes. Front Microbiol. 2016 Jun 6;7:870. doi: 10.3389/fmicb.2016.00870. eCollection 2016. PMID 27375591
- [Background] Brown RG, Marchesi JR, Lee YS, Smith A, Lehne B, Kindinger LM, Terzidou V, Holmes E, Nicholson JK, Bennett PR, MacIntyre DA. Vaginal dysbiosis increases risk of preterm fetal membrane rupture, neonatal sepsis and is exacerbated by erythromycin. BMC Med. 2018 Jan 24;16(1):9. doi: 10.1186/s12916-017-0999-x. PMID 29361936
- [Background] Chu DM, Ma J, Prince AL, Antony KM, Seferovic MD, Aagaard KM. Maturation of the infant microbiome community structure and function across multiple body sites and in relation to mode of delivery. Nat Med. 2017 Mar;23(3):314-326. doi: 10.1038/nm.4272. Epub 2017 Jan 23. PMID 28112736
- [Background] Huurre A, Kalliomaki M, Rautava S, Rinne M, Salminen S, Isolauri E. Mode of delivery - effects on gut microbiota and humoral immunity. Neonatology. 2008;93(4):236-40. doi: 10.1159/000111102. Epub 2007 Nov 16. PMID 18025796
- [Background] Mueller NT, Bakacs E, Combellick J, Grigoryan Z, Dominguez-Bello MG. The infant microbiome development: mom matters. Trends Mol Med. 2015 Feb;21(2):109-17. doi: 10.1016/j.molmed.2014.12.002. Epub 2014 Dec 11. PMID 25578246
- [Derived] Foessleitner P, Pjevac P, Granser S, Wisgrill L, Pummer L, Eckel F, Seki D, Berry D, Hausmann B, Farr A. The maternal microbiome in pregnancy, delivery, and early-stage development of neonatal microbiome after cesarean section: A prospective longitudinal study. Acta Obstet Gynecol Scand. 2024 May;103(5):832-841. doi: 10.1111/aogs.14773. Epub 2024 Jan 24. PMID 38268221